CLINICAL TRIAL: NCT04532008
Title: The ASHA Project: Pilot Study of a Depression Treatment/Economic Empowerment
Brief Title: Depression Treatment and Economic Empowerment
Acronym: ASHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Alison Karasz, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-2320
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: 48 women randomized to either intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention
- Treatment Group (Experimental): Experimental group received 12 session of group based depression treatment, a matched savings program, financial literacy training, agricultural training, and a cash transfer.
  Interventions: Behavioral: Group based treatment

INTERVENTIONS:
Behavioral: Group based treatment — 12 sessions of group based therapy that included cognitive restructuring, behavioral activation, and interpersonal therapy
  Arms: Treatment Group

SUMMARY:
This pilot study randomized 48 depressed rural Bangladeshi housewives to either intervention or control groups. The intervention groups received depression treatment and a financial empowerment intervention.

DETAILED DESCRIPTION:
This study was conducted in the rural Sirajganj region of Bangladesh. Working with the International Centre for Diarrhoeal Disease Research, Bangladesh and a local NGO, we recruited 48 depressed rural housewives for the study. Participants were randomized into intervention in control groups. The intervention groups (n=24) received 12 sessions of evidence based depression treatment, financial literacy education, agricultural training and skill building. They opened bank accounts and saved for six months. At the end of the six month period, participants who had met savings and attendance requirements received a cash transfer of approximately $186, which was used to purchase a productive asset. 22 participants purchased an agricultural animal, usually a goat; 1 financed a small retail business, and 1 leased land to grow crops for sale. Depression scores on the PHD-9 were sharply reduced. The study had 100% retention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* PHQ greater than 10
* Able to save
* Able to read and write

Exclusion Criteria:

* Not in age range PhQ below 10 Unable to contribute to savings account Illiterate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 12 months post baseline
  symptoms on the Patient Health Questionnaire (PHD-9), ranging from 0 to 27, with higher scores indicating worse outcomes

SECONDARY OUTCOMES:
Retention | Assessed at 12 Months post basline
  Percentage of participants in the intervention group completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alison Karasz, Principal Investigator — Albert Einstein College of Medicine

IPD SHARING:
Plan to Share IPD: No